CLINICAL TRIAL: NCT01334476
Title: VISN 19 MIRECC Research Database
Acronym: Repository
Status: Recruiting | Type: Observational
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lisa Brenner, Director of the VHA Rocky Mountain MIRECC, VA Eastern Colorado Health Care System
Other Study IDs: 10-0554
Record Dates: First submitted 2011-04-11; First posted 2011-04-13 (Estimated); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Demographic Data; History of Medical and Mental Health; History of Combat Experience; History of Suicide; Imaging Results
Keywords: Data Repository; Facilitate Recruitment of Participants for Ongoing and Future Research
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The VISN 19 MIRECC is involved in research concerned with suicide prevention in high risk populations (e.g., history of traumatic brain injury, post-traumatic stress disorder); Recruitment for future studies will continue with a similar focus. The aim of this protocol is for the VISN 19 MIRECC Research Database (V19-MRD), to have a data repository of participants for possible recruitment from other studies being conducted at the VISN 19 MIRECC. The VISN 19 MIRECC conducts numerous research projects under the review of COMIRB and the VA R&D.

DETAILED DESCRIPTION:
This protocol seeks to formally create the database that will store demographic data. The data will be used by VISN 19 MIRECC Investigators solely for recruitment purposes for future studies.

The repository data will include:

1. Data regarding individuals in existing study databases who have already provided permission to have their information stored and used for future recruitment into VISN 19 MIRECC research studies (specific data elements to be collected will be articulated below).
2. Data of individuals to be collected and saved to use for future recruitment into VISN 19 MIRECC research studies.

A restricted section of the V19-MRD will contain V19-MRD identification numbers and identifying data including name (first, last, middle initial), Social Security number, phone number(s) (primary and secondary), date of birth, and mailing address. A less restricted section of the V19-MRD will contain V19-MRD identification numbers, the COMIRB protocol number of the study the participant was recruited from, gender, year of birth, and criteria identifiers marked as present or absent (i.e., history of medical and mental health conditions, history of suicide - thoughts/behaviors, history of combat experience, and presence of imaging results).

The V19-MRD would enhance current research strategies by first allowing VISN 19 MIRECC Investigators an efficient method to conduct preliminary or ongoing investigations to determine if: 1) sufficient populations exist to conduct a study; or 2) potential participants meeting specific study criteria are included in the database who could be contacted regarding study participation. Second, with an approved protocol, the V19-MRD contact section of the database could be used to facilitate mailings to potential participants.

ELIGIBILITY:
Inclusion Criteria:

* Being a Patient at the Denver VA Medical Center
* 18 years or Older
* Participated in another study at the VISN 19 MIRECC

Exclusion Criteria:

* Not a Patient at the Denver VA Medical Center
* Younger than 18 years
* Never Participated on a Study Within the VISN 19 MIRECC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Receiving Medical Treatment at the Denver VA Medical Center 18 or older
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2010-06; Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Permission to contact for future studies | One time

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Brenner, PhD, Principal Investigator — VA ECHCS
Locations (2):
- United States (2):
  - VA Eastern Colorado Health Care System, Denver, Colorado
  - VHAECH Denver VA Medical Center, Denver, Colorado